CLINICAL TRIAL: NCT01275287
Title: Targeting Complement Activation in Antineutrophil Cytoplasmic Autoantibodies (ANCA)-Vasculitis
Brief Title: Targeting Complement Activation in Antineutrophil Cytoplasmic Autoantibodies (ANCA)-Vasculitis - Eculizumab
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: the study failed to enroll any patient and sponsor wished to stop.
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Alexion Pharmaceuticals, Inc. (Industry); National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-2218; P01DK058335 (NIH)
Record Dates: First submitted 2010-12-13; First posted 2011-01-12 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2016-09

CONDITIONS: Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis
Keywords: Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Complement Activation
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis | interventions — Cyclophosphamide; eculizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of care (Active Comparator): Standard of care for ANCA vasculitis treatment- depends on severity of disease and individual characteristics and medical history of each patient so this won't be described here.
  Interventions: Drug: Standard of care treatment
- Eculizumab arm (Experimental): Standard of care for ANCA vasculitis + eculizumab treatment
  Standard of care for ANCA vasculitis treatment- depends on severity of disease and individual characteristics and medical history of each patient so this won't be described here.
  Interventions: Drug: eculizumab

INTERVENTIONS:
Drug: Standard of care treatment — induction : pulse methyl prednisolone (7 mg/kg/day x3) then prednisone 1 mg/kg/day (not to exceed 60 mg/day) for 4 weeks, then taper over the following 12 weeks. Cyclophosphamide starting at 0.75 gm/m2 IV (decreased to 0.5 gm/m^2 for patients > than 70 or with estimated Glomerular Filtration Rate (eGFR) < 20 ml/min) to be titrated up to 1 gm/m^2 depending on the 2 week white blood count (WBC) nadir > 3000 cell/μL. Subsequent cyclophosphamide will be given every 4 weeks for at least 2 more doses. Once complete remission for 2 months, patient may be switched from cyclophosphamide to maintenance therapy with azathioprine 1.5-2 mg/kg/day for 6-9 months (to a total of 12 months of therapy) .
  For patients who cannot tolerate cyclophosphamide, or who have received it in large doses previously, another medication called rituximab may be used instead. However, if rituximab is indicated for the patient, he cannot participate in the study.
  Other Names: cytoxan
  Arms: Standard of care
Drug: eculizumab — In addition to conventional therapy, patients randomized to eculizumab will receive 600 mg by IV infusion over 35 minutes every 7 days for the first 4 weeks, then 900 mg by IV infusion for the fifth dose 7 days later (week 5), then 900 mg every 14 days thereafter, for a total of 9 doses (about 3 months of treatment). This dosing scheme is based on that used for the treatment of Paroxysmal Nocturnal Hemoglobinuria (PNH). The length of treatment is shorter than for PNH, based on a desire to target the addition of eculizumab to the period of maximal disease activity, while limiting the risks of infectious complications in this first pilot study.
  Other Names: Soliris
  Arms: Eculizumab arm

SUMMARY:
The purpose of this research study is to see if Eculizumab (Soliris®) can safely be used in addition to conventional therapy in patients with active ANCA (Antineutrophil Cytoplasmic Autoantibodies ) vasculitis and lead to a more rapid decrease in disease activity.

ANCA vasculitis is an inflammation of the small vessels whereby ANCA antibodies inappropriately activate one's own white blood cells (neutrophils) and cause damage to the small blood vessels.

DETAILED DESCRIPTION:
Recent laboratory studies have identified that an important pathway of inflammation called the "complement pathway" may play an important role in how Antineutrophil Cytoplasmic Autoantibodies (ANCA) cause damage to the blood vessels. Eculizumab is a monoclonal antibody that targets a key component of the complement pathway named C5, and blocks its activation.

In a mouse model of ANCA vasculitis, it has been shown that blocking C5 activation can block the development of vasculitis or greatly reduce its severity.

The researchers in this study would like to see if taking eculizumab, in addition to the drugs usually used to treat ANCA vasculitis, would be beneficial in treating ANCA vasculitis.

Currently, the conventional treatment of ANCA vasculitis consists of corticosteroids and cyclophosphamide. The corticosteroids are given as by vein (methylprednisolone) for 3 days followed by prednisone by mouth daily for about 4-5 months. Cyclophosphamide is typically given by vein every 4 weeks for at least 3 months, but sometimes longer depending on whether the vasculitis is still active or not. After the vasculitis is in remission, a maintenance treatment with azathioprine or mycophenolate mofetil may be used. For patients who cannot tolerate cyclophosphamide, or who have received it in large doses previously, another medication called rituximab may be used instead. However, patients who need rituximab or have recently been treated with rituximab cannot participate in this study.

The study drug, eculizumab, is Food and Drug Administration (FDA) approved for indications other than ANCA vasculitis. It is an investigational drug and it is NOT FDA-approved for the treatment of ANCA vasculitis.

In this study, eculizumab will be given in addition to the standard of care treatment for the patients that will be randomised to the eculizumab group.

ELIGIBILITY:
Inclusion Criteria:• Patients with active Antineutrophil Cytoplasmic Autoantibodies (ANCA) glomerulonephritis and/or small vessel vasculitis with de novo or relapsing disease (BVAS≥5).

* Patients must have a current or a history of positive ANCA by the ELISA technique.
* De novo or relapsing disease requiring immunosuppression.
* Patients must have evidence of active glomerulonephritis as evidenced by the presence of glomerular hematuria (dysmorphic Red Blood Cells (RBCs) or RBC casts) with or without an increase in serum creatinine.
* Patients will be eligible within 10 days of commencing induction therapy (i.e., they may have already received pulse methylprednisolone and first dose of cyclophosphamide).

Exclusion Criteria:• Pregnancy or lactation, or women of child bearing potential who are not willing or able to comply with 2 contraceptive methods.

* Patients with severe renal failure: creatinine > 6 mg/dL or receiving hemodialysis and/or receiving plasmapheresis therapy.
* Patients with severe pulmonary hemorrhage requiring ventilation and/or plasmapheresis therapy.
* Patients with active bacterial or viral infection.
* Absolute neutrophils count < 1000/mm^3 to minimize the risk of infections
* Hemoglobin < 8.5 g/dL
* Prior therapy with a monoclonal antibody (for example rituximab)within the previous 6 months. Peripheral CD-20 B-cells count <= 1% due to rituximab even longer than 6 months.
* Severe coexisting conditions precluding immunosuppressive therapy or conditions requiring intravenous antibiotic therapy.
* History of infection with Hepatitis B virus (HBV), Hepatitis C virus (HCV), HIV, tuberculosis or syphilis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Birmingham Vasculitis Activity Score (BVAS) | 12 weeks
  Change in disease activity as measured by BVAS at 12 weeks.

SECONDARY OUTCOMES:
Complement levels elevation | up to 52 weeks
  Evaluation of complement levels at study entry to determine which may be elevated in active disease (Bb, C3a, C3d, C3d/C3, C4d, C5a or C5b-9
Birmingham Vasculitis Activity Score(BVAS) | up to 52 weeks
  Percent of patients with a BVAS =0 at 3 months
Normalisation of complement activation | up to 52 weeks
  Normalization of complement activation at 4 weeks, 8, 12, 24, 36 and 52 weeks
Change in complement levels | from baseline to week 12
  Change in complement levels between groups from baseline to week 12
change in complement levels 2 | up to 52 weeks
  Change in these complement levels with treatment and decrease in disease activity for each patient
Birmingham Vasculitis Activity Score (BVAS) 2 | up to 52 weeks
  Mean BVAS at 24, 36 and 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Patrick H Nachman, MD, Principal Investigator — UNC Kidney Center
Locations (1):
- UNC Kidney Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
no plan too share data

REFERENCES:
- [Derived] Bala MM, Malecka-Massalska TJ, Koperny M, Zajac JF, Jarczewski JD, Szczeklik W. Anti-cytokine targeted therapies for ANCA-associated vasculitis. Cochrane Database Syst Rev. 2020 Sep 29;9(9):CD008333. doi: 10.1002/14651858.CD008333.pub2. PMID 32990324